CLINICAL TRIAL: NCT03708419
Title: Personalized Glucose Optimization Through Nutritional Intervention
Acronym: PERSON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Wageningen University and Research (Other); Top Institute Food and Nutrition (Other); Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL63768.068.17
Record Dates: First submitted 2018-04-25; First posted 2018-10-17 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Obesity; Pre-diabetic; Type 2 Diabetes Mellitus
Keywords: Insulin resistance; Personalized nutrition
MeSH Terms: conditions — Obesity; Glucose Intolerance; Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimal diet (Experimental): Participants will follow a diet for a total duration of 12 weeks, optimal for their metabolic phenotype. For participants with muscle insulin resistance (MIR) this will be a diet high in monounsaturated fatty acids, for participants with liver insulin resistance (LIR) this will be a diet high in protein and fiber and low in fat.
  Interventions: Other: Optimal diet
- Suboptimal diet (Experimental): Participants will follow a diet for a total duration of 12 weeks, suboptimal for their metabolic phenotype. For participants with liver insulin resistance (LIR) this will be a diet high in monounsaturated fatty acids, for participants with muscle insulin resistance (MIR) this will be a diet high in protein and fiber and low in fat.
  Interventions: Other: Suboptimal diet

INTERVENTIONS:
Other: Optimal diet — Based on a 7-points OGTT, participants will be classified as MIR or LIR. The hypothesized optimal diet for MIR has a moderate fat content which is high in mono- unsaturated fatty acids (HMUFA) with a macronutrient breakdown of 38 E% from fat (20% MUFA, 10% polyunsaturated fatty acids (PUFA), 8% saturated fatty acids (SFA)), 48 E% from carbohydrates (CHO, 35% complex), and 14 E% from protein (35-40% plant protein). The hypothesized optimal diet for LIR is low in fat, high in protein (LFHP) and increased fiber with a macronutrient breakdown of <28 E% from fat (10% MUFA, 10% PUFA, 8% SFA), 48 E% from CHO (35% complex), and 24 E% from protein (35-40% plant protein), and an additional supplement of 6g of soluble fiber per day. Participants wil be randomly allocated to one of the two diets.
  Arms: Optimal diet
Other: Suboptimal diet — The optimal diet for the other metabolic phenotype will be considered as "suboptimal"/ control diet. For the MIR phenotype this is the high protein, high fiber, low fat diet; for the LIR phenotype this is the high monounsaturated fatty acid diet. See the description above.
  Arms: Suboptimal diet

SUMMARY:
Maintaining well-controlled blood glucose concentrations is essential in the prevention of chronic cardiometabolic diseases. The blood glucose response to dietary and/or lifestyle patterns may vary between individuals. Insulin resistance in specific metabolic organs such as skeletal muscle, adipose tissue or the liver may underlie differential blood glucose responses.

This dietary intervention study aims to obtain insight into the metabolic and lifestyle determinants of postprandial blood glucose responses, and to establish the effect of macronutrient manipulation of a 12-week dietary intervention on blood glucose homeostasis in metabolically different subgroups an its relationship to physical and mental performance and well-being.

DETAILED DESCRIPTION:
Study design: this study is a double-blinded, randomised, controlled, parallel design dietary intervention study. The study will be conducted at Maastricht University and Wageningen University and Research, the Netherlands.

Study population: the study population will consist of 240 men and women between 40-75 years old, with a BMI 25-40 kg/m2. Participants will be either muscle insulin resistant (MIR) or liver insulin resistant (LIR), as classified by an oral glucose tolerance test (OGTT) during the screening procedure. A subgroup of 80 participants will be selected for detailed metabolic phenotyping.

Intervention: for 12 weeks, participants will receive either a diet optimal for MIR (high in mono-unsaturated fatty acids) or a diet optimal for LIR (high in protein and fiber, low in fat) with respect to changes in disposition index. Participants will be randomly allocated to one of the two diets. Detailed laboratory and daily life phenotyping will be done pre- and post intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI 25 to <40 kg/m2
* Predominantly muscle (MIR) or liver (LIR) insulin resistant
* Weight stability for at least 3 months (+/- 3 kg)

Exclusion Criteria:

Diseases

* Pre-diagnosis of type 1 or type 2 diabetes mellitus
* Renal or hepatic malfunctioning (pre-diagnosis or determined based on alanine aminotransferase (ALAT), aspartate aminotransferase (ASAT) and creatinine values)
* Gastrointestinal diseases or abdominal surgery (allowed i.e.: appendectomy, cholecystectomy)
* Food allergies, intolerances (including gluten/lactose intolerance) and/or dietary restrictions interfering with the study (including special diets, vegetarians and eating disorders)
* Cardiovascular diseases (e.g. heart failure) or cancer (e.g. non-invasive skin cancer allowed)
* High blood pressure (untreated >160/100 mmHg, drug-regulated >140/90 mmHg)
* Diseases affecting glucose and/or lipid metabolism (e.g. pheochromocytoma, Cushing's syndrome, acromegaly)
* Anemia defined as hemoglobin (Hb) men <8.5 and women <7.5 mmol/l
* Diseases with a life expectation shorter than 5 years
* Major mental disorders
* Drug treated thyroid diseases (well substituted hypothyroidism is allowed inclusion)
* Other physical/mental conditions that could interfere with study outcomes

Medication

* Medication known to interfere with study outcomes (e.g. peroxisome proliferator-activated receptor-α (PPAR-α) or PPAR-γ agonists (fibrates), sulfonylureas, biguanides, α-glucosidase inhibitors, thiazolidinediones, repaglinide, nateglinide and insulin, chronic use of NSAIDs)
* Use of anticoagulants
* Use of antidepressants (stable use ≥ 3 months prior to and during the study is allowed)
* Use of statins (stable use ≥ months prior to and during study allowed)
* Use of β-blockers (only for the extensive phenotyping participants)
* Chronic corticosteroids treatment (>7 consecutive days of treatment)
* Use of antibiotics within 3 months prior to the study

Lifestyle

* Participation in regular sports activities (>4 hours per week)
* Having a restricted dietary pattern interfering with the study diets (e.g. vegan or Atkins diet)
* Plans to lose weight
* Abuse of alcohol (alcohol consumption >14 units/week) and/or drugs (cannabis included)
* Not willing to limit alcohol consumption to 7 drinks per week
* Regular smoking (including use of e-cigarettes)
* Use of strong vitamins or dietary supplements (e.g. pre- or probiotics) expected to interfere with the study outcomes

Other

* Pregnant or lactating women who are planning to become pregnant
* Inability to comply with the study diet
* Blood donation within the last 3 months
* Participation in possibly interfering studies within the last 3 months
* Inability to understand study information and/or communicate with staff
* Unwillingness to be randomized or sign informed consent
* Unwillingness to save data for 15 years

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2021-11-29 (Actual); Study Completion 2021-11-29 (Actual)

PRIMARY OUTCOMES:
Disposition index | Change from baseline at week 12 dietary intervention
  The primary objective of this study is to establish the effect of a metabolically targeted, optimal versus suboptimal macronutrient manipulated 12-week dietary intervention on the change in disposition index, a composite marker of first phase insulin secretion and insulin sensitivity during a 2-hour 7-points oral glucose tolerance test (OGTT). Disposition index will be calculated as follows: [Insulin sensitivity index (ISI) * (AUC30 min insulin / AUC30 min glucose)], where AUC30 min is the area under the curve between 0 and 30 minutes of the OGTT for insulin (pmol/l) and glucose (mmol/l), respectively, and ISI is defined as: [10,000 ÷ square root of (fasting plasma glucose (mmol/l) x fasting insulin (pmol/l)) x (mean glucose (mmol/l) x mean insulin (pmol/l))]. Higher values represent a higher insulin sensitivity.

SECONDARY OUTCOMES:
Mean 24h glucose concentrations | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. The mean 24h glucose concentrations will be measured continuously with the iPro2 device and Enlite Glucose Sensor (Medtronic) and expressed as mmol/L.
Glucose incremental area under the curve (iAUC) | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. The iAUC will be calculated using the trapezoid rule from data obtained from the iPro2 device and Enlite Glucose Sensor (Medtronic). The iAUC provides a summary measure of the net increase in glucose levels above the fasting level during a 24-hour period and is expressed as mmol/min/L.
The frequency and duration of hypo- and hyperglycemia | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. The frequency and duration of hypo- and hyperinsulinemia will be monitored using the iPro2 device and Enlite Glucose Sensor (Medtronic) and is defined as a glucose level of ≥10.0 mmol/l for hyperglycemia, whilst hypoglycemia will be defined as a glucose concentration ≤3.9 mmol/l.
Glucose tolerance | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Determined by 2-hour glucose values (mmol/L) during an oral glucose tolerance test.
Muscle insulin sensitivity | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Determined during a 2-hour, 7-points oral glucose tolerance test. The muscle insulin sensitivity index (MISI) will be calculated as follows: MISI (mmol/l/min/pmol/l) = (dG/dt) / mean plasma insulin concentration (pmol/l) during OGTT. Here, dG/dt is the rate of decay of plasma glucose concentration (mmol/L) during the OGTT, calculated as the slope of the least square fit to the decline in plasma glucose concentration from peak to nadir. Higher values represent higher muscle insulin sensitivity.
Hepatic insulin sensitivity | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Determined during a 2-hour, 7-points oral glucose tolerance test. The hepatic insulin resistance index (HIRI) will be calculated using the square root of the product of the area under curves (AUCs) for glucose and insulin during the first 30 min of the OGTT - i.e., square root (glucose0-30 [AUC in mmol/l·h] · insulin 0-30 [AUC in pmol/l·h). Higher IR values represent lower hepatic insulin sensitivity.
Insulin sensitivity | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Glucose infusion rate (mg/kg/min) during a 2-step hyper-insulinemic euglycemic clamp as golden standard method.
Body composition | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Body composition will be determined by using a dual-energy X-ray absorptiometry scan (DXA).
Waist circumference | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Waist circumferences in centimeters.
Hip circumferences | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Hip circumferences in centimeters.
Body fat distribution | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Magnetic Resonance Imaging (MRI)(UM) and Magnetic resonance spectroscopy (1H-MRS)(WUR) measurements will be included to quantify both subcutaneous and visceral fat depots, and ectopic fat deposition (e.g. in liver and muscle).
Blood pressure | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Systolic and diastolic blood pressure in mmHg.
Fasting circulating metabolic markers | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Fasting circulating metabolic markers include: glucose, insulin, hemoglobin A1c (HbA1c), triacylglycerol, free glycerol, free fatty acids (FFA), lactate, high density lipoprotein (HDL), total cholesterol, short chain fatty acids (SCFA), bile acids, glucagon-like peptide-1 (GLP-1), peptide YY (PYY).
Fasting blood lipid spectrum | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Metabolomics will be used to determine the fasting blood lipid spectrum.
Postprandial circulating metabolic markers | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Postprandial circulating metabolic markers will be determined during a high-fat mixed-meal test and include: glucose, insulin, triacylglycerol, free glycerol, free fatty acids (FFA), lactate, high density lipoprotein (HDL), total cholesterol, short chain fatty acids (SCFA), bile acids, glucagon-like peptide-1 (GLP-1), peptide YY (PYY).
Energy expenditure | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Fasting and insulin-stimulated energy expenditure will be determined by indirect calorimetry during a 2-step hyperinsulinemic-euglycemic clamp.
Substrate oxidation | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Fasting and insulin-stimulated substrate oxidation will be determined by indirect calorimetry during a 2-step hyperinsulinemic-euglycemic clamp.
Fecal microbiota composition | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Fecal samples to be used for analysing microbiota composition will be collected.
Oral microbiota composition | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Saliva samples to be used for analysing microbiota composition will be collected.
Self-reported perceived stress | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Perceived stress will be assessed using a 10-item perceived stress scale (PSS-10). Items will be scored based on a 5-point Likert scale, with higher scores representing higher perceived stress levels.
Self-reported self efficacy in physical activity | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Self efficacy in physical activity will be assessed using Likert scales, determining an individual's ability to achieve performing physical activity.
Self-reported sleep behaviour | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Sleep behaviour will be assessed using the Munich Chronotype Questionnaire (MCTQ).
Self-reported sleep quality over a 1 month period | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Sleeping quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI).
Self-reported daytime sleepiness | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Daytime sleepiness is assessed using the 8-item Epworth Sleepiness Scale (ESS). Items will be scored on a scale of 0-3, with a higher score representing a higher probability of falling asleep.
Self-reported fatigue | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Self-reported fatigue will be assessed using the Chalder Fatigue Scale.
Self-reported sedentary behaviour | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Sedentary behaviour will be assessed using the sedentary behaviour questionnaire (AQUAA).
Self-reported physical activity | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Self-reported physical activity will be assessed using the physical activity questionnaire (Baecke).
Self-reported eating rate | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Self-reported eating rate will be assessed using the eating rate index.
Self-reported intestinal health | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Self-reported intestinal health will be assessed using an intestinal health questionnaire and the Bristol Stool Chart.
Self-reported quality of life | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Self-reported quality of life will be assessed using the 36-Item Short Form Health Survey (SF-36). Higher scores represent less disability.
Physical activity patterns | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Physical activity patterns will be monitored continuously with the ActivPAL3 device.
Cognitive performance | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Cognitive function will be assessed using the Cambridge Neuropsychological Test Automated Battery.
Subcutaneous adipose tissue biopsy | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Subcutaneous adipose tissue biopsies will be taken for histology and gene and protein expression analysis.
Skeletal muscle biopsy | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Skeletal muscle biopsies will be taken for histology and gene and protein expression analysis.
Advanced glycation end-product (AGE) accumulation | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. AGE accumulation will be measured by skin autofluorescence using an AGE reader (Diagnoptics)
Fasting immune metabolism (PBMCs) | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Assessment of PBMCs as measure of fasting immune metabolism
Carotid artery reactivity | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Assessment of (peripheral) vascular function by carotid artery reactivity (CAR) in response to a cold pressor test.
Food preferences | Change from baseline at week 12 dietary intervention
  Optimal versus suboptimal diet. Food preferences will be assessed by using the computer-based Macronutrient and Taste Preference Ranking Task (MTPRT).
Intervention effects on all above outcomes within the LIR and MIR group. | Change from baseline at week 12 dietary intervention
  In contrast to the other outcomes, the intervention effect within the MIR and LIR group will be analysed for all above mentioned outcomes (as compared to an analysis of optimal versus the suboptimal diet). MIR and LIR are two measures of insulin resistance, in primarily the muscle and liver, respectively. MIR and LIR can be modelled from an OGTT, as described above. Thus, for each of the outcomes described above, their change following 12 weeks of dietary intervention will be compared between the two metabolic phenotypes, MIR and LIR.
DNA analysis | Baseline
  Buffy coats will be collected for DNA analysis, pre-intervention only.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen E Blaak, Prof., Principal Investigator — Maastricht University
Locations (2):
- Netherlands (2):
  - Department of Human Biology, Maastricht University Medical Centre, Maastricht
  - Wageningen University and Research, Wageningen

REFERENCES:
- [Derived] Jardon KM, Umanets A, Gijbels A, Trouwborst I, Hul GB, Siebelink E, Vliex LMM, Bastings JJAJ, Argamasilla R, Chenal E, Venema K, Afman LA, Goossens GH, Blaak EE. Distinct gut microbiota and metabolome features of tissue-specific insulin resistance in overweight and obesity. Gut Microbes. 2025 Dec;17(1):2501185. doi: 10.1080/19490976.2025.2501185. Epub 2025 May 7. PMID 40336254
- [Derived] Gijbels A, Jardon KM, Trouwborst I, Manusama KC, Goossens GH, Blaak EE, Feskens EJ, Afman LA. Fasting and postprandial plasma metabolite responses to a 12-wk dietary intervention in tissue-specific insulin resistance: a secondary analysis of the PERSonalized glucose Optimization through Nutritional intervention (PERSON) randomized trial. Am J Clin Nutr. 2024 Aug;120(2):347-359. doi: 10.1016/j.ajcnut.2024.05.027. Epub 2024 Jun 6. PMID 38851634
- [Derived] Trouwborst I, Jardon KM, Gijbels A, Hul G, Feskens EJM, Afman LA, Linge J, Goossens GH, Blaak EE. Body composition and body fat distribution in tissue-specific insulin resistance and in response to a 12-week isocaloric dietary macronutrient intervention. Nutr Metab (Lond). 2024 Apr 9;21(1):20. doi: 10.1186/s12986-024-00795-y. PMID 38594756
- [Derived] Trouwborst I, Gijbels A, Jardon KM, Siebelink E, Hul GB, Wanders L, Erdos B, Peter S, Singh-Povel CM, de Vogel-van den Bosch J, Adriaens ME, Arts ICW, Thijssen DHJ, Feskens EJM, Goossens GH, Afman LA, Blaak EE. Cardiometabolic health improvements upon dietary intervention are driven by tissue-specific insulin resistance phenotype: A precision nutrition trial. Cell Metab. 2023 Jan 3;35(1):71-83.e5. doi: 10.1016/j.cmet.2022.12.002. PMID 36599304
- [Derived] Gijbels A, Trouwborst I, Jardon KM, Hul GB, Siebelink E, Bowser SM, Yildiz D, Wanders L, Erdos B, Thijssen DHJ, Feskens EJM, Goossens GH, Afman LA, Blaak EE. The PERSonalized Glucose Optimization Through Nutritional Intervention (PERSON) Study: Rationale, Design and Preliminary Screening Results. Front Nutr. 2021 Jun 30;8:694568. doi: 10.3389/fnut.2021.694568. eCollection 2021. PMID 34277687